CLINICAL TRIAL: NCT00259922
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Phase 3 Study to Evaluate the Efficacy and Safety of Alvimopan 0.5mg Once Daily and 0.5mg Twice Daily for 12 Weeks for the Treatment of Opioid-Induced Bowel Dysfunction in Adults Taking Opioid Therapy for Persistent Non-Cancer Pain
Brief Title: Alvimopan For The Treatment Of Constipation Due To Opioids Being Taken For Persistent Non-Cancer Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SB-767905/013
Record Dates: First submitted 2005-11-29; First posted 2005-12-01 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2009-09

CONDITIONS: Bowel Dysfunction; Constipation
Keywords: constipation; gastrointestinal; opioids; pain; non-cancer pain; opioid-induced; bowel dysfunction
MeSH Terms: conditions — Intestinal Diseases; Constipation; Pain | interventions — alvimopan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Alvimopan 0.5 mg once daily (Experimental): 0.5 mg once daily (QD)
  Interventions: Drug: Alvimopan
- Alvimopan 0.5 mg twice daily (Experimental): 0.5 mg twice daily (BID)
  Interventions: Drug: Alviompan

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: Placebo
Drug: Alvimopan — 0.5 mg QD
  Other Names: Entereg
  Arms: Alvimopan 0.5 mg once daily
Drug: Alviompan — 0.5 mg BID
  Other Names: Entereg
  Arms: Alvimopan 0.5 mg twice daily

SUMMARY:
Adults who are taking opioid therapy for persistent non-cancer pain and have resulting opioid-induced bowel dysfunction (OBD) will be randomized (1:1:1) to one of 2 alvimopan arms, or to placebo. The primary objective of this phase 3 confirmatory study is to compare alvimopan with placebo for efficacy in the treatment of OBD. The primary efficacy endpoint is based on frequency of bowel movements. Subjects will be required to: (1) track their bowel movements and other bowel symptoms and (2) attend 6 clinic visits over 4 months.

ELIGIBILITY:
Inclusion criteria:

* Consented to participate in this study.
* Taking opioid therapy for persistent non-cancer pain.
* Has bowel dysfunction mainly due to opioids.
* Has bowel dysfunction since starting opioids as defined by infrequent bowel movements and additional bowel-related symptoms.
* Willing to discontinue laxative therapy (will be provided study-specific standardized laxative if needed).
* Willing to report daily bowel symptoms.

Exclusion criteria:

* Pregnant, lactating, or planning to become pregnant.
* Not ambulatory.
* Participated in another trial with an investigational drug in the past 30 days.
* Taking opioids for the management of drug addiction or cancer-related pain.
* Severe constipation whereby the subject is at immediate risk of developing serious complications of constipation.
* Gastrointestinal or pelvic disorders known to affect bowel transit, produce gastrointestinal (GI) obstruction, or contribute to bowel dysfunction.
* HIV-infected, has active hepatitis, or has ever been infected with hepatitis C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 485 (Actual)
Dates: Start 2005-08; Primary Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
To compare alvimopan with placebo for efficacy in the treatment of OBD

SECONDARY OUTCOMES:
Safety and tolerability, quality of life, pharmacogenetics (dependent on results from other data)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (170):
- United States (107):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Huntsville, Alabama
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Northport, Alabama
  - GSK Investigational Site, Mesa, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Tempe, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Los Gatos, California
  - GSK Investigational Site, Northridge, California
  - GSK Investigational Site, Orange, California
  - GSK Investigational Site, Palm Springs, California
  - GSK Investigational Site, Pasadena, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, San Rafael, California
  - GSK Investigational Site, Santa Ana, California
  - GSK Investigational Site, Stamford, Connecticut
  - GSK Investigational Site, Waterbury, Connecticut
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Chiefland, Florida
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Deerfield Beach, Florida
  - GSK Investigational Site, Destin, Florida
  - GSK Investigational Site, Fort Myers, Florida
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Largo, Florida
  - GSK Investigational Site, Margate, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Ocala, Florida
  - GSK Investigational Site, Ormond Beach, Florida
  - GSK Investigational Site, Saint Cloud, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Winterhaven, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Cumming, Georgia
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Stockbridge, Georgia
  - GSK Investigational Site, Meridian, Idaho
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Libertyville, Illinois
  - GSK Investigational Site, Oak Forest, Illinois
  - GSK Investigational Site, Oakbrook Terrace, Illinois
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Sunset, Louisiana
  - GSK Investigational Site, Pasadena, Maryland
  - GSK Investigational Site, Rockville, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Brockton, Massachusetts
  - GSK Investigational Site, Wellesley Hills, Massachusetts
  - GSK Investigational Site, Portage, Michigan
  - GSK Investigational Site, Waterford, Michigan
  - GSK Investigational Site, Olive Branch, Mississippi
  - GSK Investigational Site, Independence, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Missoula, Montana
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Dover, New Hampshire
  - GSK Investigational Site, Blackwood, New Jersey
  - GSK Investigational Site, Egg Harbor, New Jersey
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Mineola, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Asheville, North Carolina
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Hickory, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Centerville, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Perrysburg, Ohio
  - GSK Investigational Site, Eugene, Oregon
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Salem, Oregon
  - GSK Investigational Site, Levittown, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Reading, Pennsylvania
  - GSK Investigational Site, Cranston, Rhode Island
  - GSK Investigational Site, Greer, South Carolina
  - GSK Investigational Site, Kingsport, Tennessee
  - GSK Investigational Site, New Tazewell, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Corpus Christi, Texas
  - GSK Investigational Site, Galveston, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Richardson, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Tacoma, Washington
  - GSK Investigational Site, Yakima, Washington
  - GSK Investigational Site, Charleston, West Virginia
  - GSK Investigational Site, La Crosse, Wisconsin
- Australia (12):
  - GSK Investigational Site, Broadmeadow, New South Wales
  - GSK Investigational Site, Newcastle, New South Wales
  - GSK Investigational Site, St Leonards, New South Wales
  - GSK Investigational Site, Carina Heights, Queensland
  - GSK Investigational Site, Kippa-Ring, Queensland
  - GSK Investigational Site, Bedford Park, South Australia
  - GSK Investigational Site, Port Lincoln, South Australia
  - GSK Investigational Site, Toorak Gardens, South Australia
  - GSK Investigational Site, Box Hill, Victoria
  - GSK Investigational Site, Carlton, Victoria
  - GSK Investigational Site, Fremantle, Western Australia
  - GSK Investigational Site, Nedlands, Western Australia
- Canada (11):
  - GSK Investigational Site, Coquitlam, British Columbia
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Moncton, New Brunswick
  - GSK Investigational Site, St. John's, Newfoundland and Labrador
  - GSK Investigational Site, Greater Sudbury, Ontario
  - GSK Investigational Site, Mississauga, Ontario
  - GSK Investigational Site, North Bay, Ontario
  - GSK Investigational Site, North York, Ontario
  - GSK Investigational Site, Bonaventure, Quebec
  - GSK Investigational Site, Saint Romuald, Quebec
  - GSK Investigational Site, Trois-Rivières, Quebec
- France (4):
  - GSK Investigational Site, Boulogne
  - GSK Investigational Site, Grenoble
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Paris
- Hungary (3):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Csongrád
  - GSK Investigational Site, Heves
- Netherlands (5):
  - GSK Investigational Site, Alkmaar
  - GSK Investigational Site, Breda
  - GSK Investigational Site, Roosendaal
  - GSK Investigational Site, Rotterdam
  - GSK Investigational Site, Utrecht
- New Zealand (3):
  - GSK Investigational Site, Christchurch
  - GSK Investigational Site, Hamilton
  - GSK Investigational Site, Tauranga
- Norway (4):
  - GSK Investigational Site, Oslo
  - GSK Investigational Site, Paradis
  - GSK Investigational Site, Rådahl
  - GSK Investigational Site, Skien
- South Africa (8):
  - GSK Investigational Site, Athlone, Cape Town
  - GSK Investigational Site, Erasmuskloof, Pretoria
  - GSK Investigational Site, Fourways, Johannesburg
  - GSK Investigational Site, Kempton Park
  - GSK Investigational Site, Kenilworth, Cape Town
  - GSK Investigational Site, Lynnwood, Pretoria
  - GSK Investigational Site, Tygervalley
  - GSK Investigational Site, Westridge, Mitchells Plain
- Spain (7):
  - GSK Investigational Site, Alcorcón
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Ferrol
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Valencia
- Sweden (4):
  - GSK Investigational Site, Jönköping
  - GSK Investigational Site, Karlstad
  - GSK Investigational Site, Linköping
  - GSK Investigational Site, Stockholm
- Switzerland (2):
  - GSK Investigational Site, Bern
  - GSK Investigational Site, Nottwil

REFERENCES:
- [Result] Irving G, Penzes J, Ramjattan B, Cousins M, Rauck R, Spierings EL, Kleoudis CS, Snidow JW, Pierce A, Wurzelmann J, Mortensen ER. A randomized, placebo-controlled phase 3 trial (Study SB-767905/013) of alvimopan for opioid-induced bowel dysfunction in patients with non-cancer pain. J Pain. 2011 Feb;12(2):175-84. doi: 10.1016/j.jpain.2010.06.013. PMID 21292168